CLINICAL TRIAL: NCT00682071
Title: Abdominal Versus Transvaginal Ultrasound Guided Embryo Transfer: Results of a Randomized Clinical Trial
Brief Title: Ultrasound Guided Embryo Transfer: Abdominal Versus Transvaginal, a RCT
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-311; IRB# 2003-311 (UW); HSC# 2003-311 (UW); Grant: OB/GYN R&D; Funding # 133-FZ71
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-05

CONDITIONS: Infertility; in Vitro Fertilization
Keywords: Ultrasound-guided; embryo transfer; in-vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: transabdominal ultrasound (TAS) guided embryo transfer
- 2: transvaginal ultrasound (TVS) guided embryo transfer

SUMMARY:
Ultrasound (US) guided embryo transfer (ET) appears to improve pregnancy outcomes in IVF-ET. Most reports are done using a transabdominal (TAS) approach, in contrast to a transvaginal ultrasound (TVS) which does not require a full bladder. We sought to determine if either approach was better with respect to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing assisted reproductive cycles including autologous IVF, oocyte donation, and frozen embryo transfer (FET) cycles

Exclusion Criteria:

- Cases of severe ovarian hyper-stimulation requiring embryo cryopreservation and gestational surrogate cycles

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing assisted reproductive cycles at the University of Wisconsin REI Program
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2003-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
pregnancy rates for TAS and TVS ultrasound-guided ET groups | August 2003 to June 2007

SECONDARY OUTCOMES:
Length of time required for embryo transfer | August 2003 to June 2007
differences between transferring physicians | August 2003 to June 2007
multiple pregnancies | August 2003 to June 2007
ectopic pregnancy rates | August 2003 to June 2007

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Lindheim, MD, MMM, Principal Investigator — Fertility Specialists Medical Group